CLINICAL TRIAL: NCT03127449
Title: Multiple-Centered Study of AST2818 in Patients With Advanced Non-small Cell Lung Cancer With EGFR Mutations
Brief Title: AST2818 in Advanced Non-Small Cell Lung Cancer With EGFR Mutations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Indications have been approved for marketing
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170405
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Advanced NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alflutinib (Experimental): patients take Alflutinib orally once per day at different dose
  Interventions: Drug: Alflutinib

INTERVENTIONS:
Drug: Alflutinib — patients take Alflutinib orally once per day at different dose
  Other Names: AST2818

SUMMARY:
This study is conducted to assess the safety, tolerability and preliminary efficacy of AST2818 in patients with advanced Non Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged older than 18 years.
* Histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC.
* Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI e.g. gefitinib or erlotinib or Afatinib, or Icotinib (Third EGFR TKI are not included). In addition other lines of therapy may have been given.
* Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including at least one of G719X, exon 19 deletion, L858R, L861Q mutation)
* Documented evidence of definitely EGFR T790M+ state in the tumor tissue after disease progression on the most recent treatment regimen (irrespective of whether this is EGFR TKI or chemotherapy).
* ECOG performance status of 0 to 2. Life expectancy of at least 12 weeks.
* At least one measurable disease by CT or PET-CT or MRI, according to RECIST Version 1.1.
* Organ function must meet the following requirements：Absolute neutrophil count >= 1.5 x 109/L, Platelet count >= 75 x 109/L, Haemoglobin >= 90 g/L；Alanine aminotransferase/Aspartate aminotransferase <= 2.5 times the upper limit of normal if no demonstrable liver metastases or <= 5 times in the presence of liver metastases；Total bilirubin <= 1.5 times ULN if no liver metastases or <= 3 times ULN in the presence of liver metastases or liver metastases；Creatinine <=1.5 times ULN concurrent with creatinine clearance >= 50 ml/min (measured or calculated by Cockcroft and Gault equation); Females should not be in lactation period and must have a negative pregnancy test prior to start of dosing; During the whole treatment,all patients should be in the entire 3 months during and after the treatment, repeated barrier precautions
* Signed consent on an Independent Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation.

Exclusion Criteria:

* Any cytotoxic chemotherapy from a previous treatment regimen or clinical study within 21 days，Any Target cancer drug from a previous treatment regimen or clinical study within 14 days, or less than approximately 5x half-life of the first dose of study treatment；The third EGFR-TKI from a previous treatment regimen or clinical study (ie, AZD9291, CO-1686, HM61713, ASP8273, EGF816, avitinib,
* Taking (or cannot stop taking 1 week before the first dose receiving) strong inhibitor of CYP3A4 or antitumor herb.
* Unrecovered toxic reaction due to former therapy existed, with over 1 grade of CTCAE (except alopecia) or 2 grade if ever applied DDP curing related neuropathy.
* Spinal compression, or brain metastasis exhibiting symptoms but untreated (except those exhibit no symptom with stable condition and do not apply corticosteroids for 4 weeks before the trail initiating)
* Any evidence showing severe or inadequate controlled systemic disease. For example patients with inadequate controlled hypertension considered not suitable for the trail or would affect the compliance towards the protocol, with active hemorrhagic tendency, with active infection such as HBV (HBV-DNA≥1000cps/ml), with HCV, with HIV et al (except for HBV carrier those the researcher considered meet the criterion).
* Any condition affecting the drug taking, or significantly affecting the absorption or the pharmacokinetic parameters, include any kind of uncontrollable nausea or vomit, chronic gastroenteropathy, disability in swallowing, and history of gastrointestinal resection or surgery.
* Any condition meet the following cardiac standard: ECG show a QTc>470 msec under resting state (Repeat in 48 hours when a first abnormal discovered, take mean of the two measurements). All kinds of abnormal in cardiac rhythm, conduction and resting ECG profile with clinical significance, for example complete left bundle branch block, 2 or 3 grade of conduction block and a PR interval>250 msec. Any possible factors increasing the risk of QTc extending or leading to arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, any first degree relative suffered from long QT syndrome or undertook unexplained sudden death before 40 years old, or taking any drug leading to a longer QTc.
* Any history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonia require steroid therapy or active interstitial lung disease with clinical evidence during recruiting.
* Patients with other factors the researchers considered not suitable for the trail (for example, patients those who not willing to follow the procedure, limitation or requirements, who once experienced bone marrow allotransplantation, who have other kinds of malignant tumor coexisted or who showed allergic to the active ingredients or inactive adjuvant of the investigational drug, as well as drugs with similar chemical structure or in the same class).
* Confirmed mutation of EGFR 20 exon insertion at anytime after the first diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks.
  Evaluation of objective response rate assessed by RECIST 1.1

SECONDARY OUTCOMES:
Duration of response of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks.
  Duration of response assessed by RECIST 1.1
Progression free survival of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival
Clinical benefit rate of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks.
  Clinical benefit rate was calculated by adding up complete remission, partial remission and stabilization of disease assessed by RECIST 1.1
Disease control rate of Alflutinib | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression or withdrawal from study, whichever came first, assessed up to 52 weeks.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate disease control rate
Incidence and Severity of Treatment-Emergent Adverse Events | Adverse events will be collected from baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, ophthalmic examinations, RECIST1.1, and NCI CTCAE v4.03
Steady state Maximum Plasma Concentration [Cmax] of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  Cmax of Alflutinib and 2 metabolites at steady state following multiple doses
Steady state peak plasma time [tmax] of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  tmax of Alflutinib and 2 metabolites at steady state following multiple doses.
Steady state Cmin (Minimum Plasma Concentration) of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  Cmin of Alflutinib and 2 metabolites at steady state following multiple doses.
Steady state area under the plasma concentration versus time curve [AUC] of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  AUC of Alflutinib and 2 metabolites at steady state following multiple doses.
Steady state clearance of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  Clearance of Alflutinib and 2 metabolites at steady state following multiple doses.
Accumulation ratio of multiple doses Alflutinib and 2 metabolites | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 1, 8, 15. Cycle 2 D1- pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose)
  Accumulation ratio of Alflutinib and 2 metabolites following multiple doses.

CONTACTS AND LOCATIONS:
Locations (1):
- cancer hospital Chinese academy of medical sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Zhang S, Hu X, Feng J, Ma Z, Zhou J, Yang N, Wu L, Liao W, Zhong D, Han X, Wang Z, Zhang X, Qin S, Ying K, Feng J, Fang J, Liu L, Jiang Y. Safety, Clinical Activity, and Pharmacokinetics of Alflutinib (AST2818) in Patients With Advanced NSCLC With EGFR T790M Mutation. J Thorac Oncol. 2020 Jun;15(6):1015-1026. doi: 10.1016/j.jtho.2020.01.010. Epub 2020 Jan 30. PMID 32007598